CLINICAL TRIAL: NCT05676307
Title: ETIOLOGICAL FACTORS AND EFFECT OF VESTIBULAR REHABILITATION ON BILATERAL VESTIBULAR HYPOFUNCTION
Brief Title: Vestibular Rehabilitaion in Bilateral Vestibular Hypofunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gedik University (Other)
Responsible Party: Principal Investigator, Gonul ERTUNC GULCELIK, Asst. Prof., Istanbul Gedik University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31207858
Record Dates: First submitted 2022-12-02; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Bilateral Vestibular Loss; Vestibular Rehabilitation
MeSH Terms: conditions — Bilateral Vestibulopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral Vestibular Hypofunction (Experimental): Vestibular Rehabilitation in Bilateral Vestibular Hypofunction
  Interventions: Behavioral: Vestibular Rehabilitation

INTERVENTIONS:
Behavioral: Vestibular Rehabilitation — Cawthorne Cooksey Based Vestibular Rehabilitation Exercises (Oculomotor exercise, Vestibulo-ocular Exercise, posture exercise, balance training, etc)

SUMMARY:
The purpose of this study is to determine the etiological factors that constitute bilateral vestibular hypofunction and to investigate the effect of vestibular rehabilitation in these patients.

The Caloric test and Video Head Impulse test were applied to evaluate the vestibular hypofunction picture of the patients who applied to Clinic with complaints of vertigo, dizziness and imbalance. Among these patients with BVH, those with vestibular symptoms, imbalance complaints and limited daily living activities were included in rehabilitation. In order to investigate the effectiveness of rehabilitation, oculomotor functions were evaluated using Simulation Of Vestibulo-ocular Reflex Exercises (SVORE) System, balance assessment was done with timed balance tests and quality of life assessment was performed with Dizziness Handicap Inventory.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-70 years of age with bilateral vestibular hypofunction and peripheral vestibulopathy

Exclusion Criteria:

* Patients with unilateral vestibular hypofunction, cerebellar lesion, and cognitive problems were excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-10-23 (Actual); Study Completion 2022-11-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of Oculomotor Activity (Saccade Frequency Level) | 8 week
  Oculomotor Function Level was evaluated with Simulation Of Vestibulo-ocular Reflex Exercises (SVORE) System. The name of this web-based system that supports VOR wient in the evaluation part of the vestibular software.sth oculomotor and optokinetic stimuli is Simulation of Vestibulo-Ocular Reflex Exercises (SVORE). This system includes Assessment and Rehabilitation departments. The maximum saccade frequency levels were determined with the measurements. For the evaluation of saccade eye movement, patient will be asked to focus on the objects on the screen.
Quality of Life Assesment | 8 weeks
  The level of quality of life was evaluated with Dizziness Handicap inventory.The Dizziness Handicap Inventory (DHI), which evaluates the quality of life in vestibular diseases, was used in the study. This 25-item scale determines the emotional and functional outcomes of patients in vestibular system diseases as well as aggravating factors related to dizziness and impaired balance.
Static Balance Tests | 8 weeks
  To evaluate the static balance of the patients; Length of standing in romberg, semitandem, tandem, standing on one leg, eyes open-closed positions were recorded in seconds with a stopwatch.
Evaluation of Oculomotor Activity (Pursuit Frequency Level) | 8 weeks
  Oculomotor Function Level was evaluated with Simulation Of Vestibulo-ocular Reflex Exercises (SVORE) System. The name of this web-based system that supports VOR wient in the evaluation part of the vestibular software.sth oculomotor and optokinetic stimuli is Simulation of Vestibulo-Ocular Reflex Exercises (SVORE). This system includes Assessment and Rehabilitation departments. The maximum pursuit frequency levels were determined with the measurements.For the evaluation of pursuit eye movement, patient will be asked to focus continuely on the objects on the screen.

CONTACTS AND LOCATIONS:
Locations (1):
- Gönül Ertunç Gülçelik, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No